CLINICAL TRIAL: NCT01344863
Title: A Randomized, Open-label, 2-arm, Parallel Group, Single Dose, Multi-center Study in Healthy Male Subjects to Investigate the Comparability of Pharmacokinetics of Trastuzumab Administered Subcutaneously as the Trastuzumab/rHuPH20 Formulation Using a Handheld Syringe or Using the Proprietary Single-use Injection Device (SID)
Brief Title: A Study of Administration of Trastuzumab (Herceptin) by a Single-use Injection Device Versus a Handheld Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO25532
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Trastuzumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: trastuzumab [Herceptin]
- 2 (Active Comparator)
  Interventions: Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: trastuzumab [Herceptin] — 600 mg subcutaneously using a single-use injection device on Day 1
  Arms: 1
Drug: trastuzumab [Herceptin] — 600 mg subcutaneously using a handheld syringe on Day 1
  Arms: 2

SUMMARY:
This randomized, open-label, parallel, 2-arm, multicenter study will compare the administration of Herceptin (trastuzumab) with a single-use injection device versus a handheld syringe in healthy male volunteers. The volunteers will receive a single dose of 600 mg Herceptin. The anticipated time of the study is 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male patients, 18 to 45 years of age, inclusive
* No history of hypersensitivity or allergic reactions following drug administration
* No history of clinically significant or clinically relevant cardiac condition
* No history of previous anticancer treatment
* Body mass index (BMI) between 18-32 kg/m2, inclusive

Exclusion Criteria:

* Positive test result for drugs of abuse
* Positive test result for hepatitis B, hepatitis C, or HIV 1 or 2
* Systolic blood pressure greater than 140 mmHG or less than 90 mmHG, or diastolic blood pressure greater than 90 mmHG or less than 50 mmHG
* Clinically significant abnormal laboratory values

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration curve of trastuzumab | 21 days
Maximum observed plasma concentration of trastuzumab | 21 days

SECONDARY OUTCOMES:
Plasma concentration of trastuzumab | Day 21
Safety: Incidence of adverse events | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- New Zealand (2):
  - Christchurch
  - Grafton

REFERENCES:
- [Derived] Wynne CJ, Ellis-Pegler RB, Waaka DS, Schwabe C, Lehle M, Heinzmann D, Mangat R, Li C, Dick AE, Cranshaw NA, Lum BL. Comparative pharmacokinetics of subcutaneous trastuzumab administered via handheld syringe or proprietary single-use injection device in healthy males. Cancer Chemother Pharmacol. 2013 Nov;72(5):1079-87. doi: 10.1007/s00280-013-2273-z. Epub 2013 Sep 22. PMID 24057039